CLINICAL TRIAL: NCT02300337
Title: Comparative Study of the Tightness of the Laryngeal Tube Under Mechanical Ventilation Before and After Reduction of Cuff Pressure on 60cmH₂O, 50cmH₂O, 40cmH₂O or 30cmH₂O
Brief Title: Comparison of Reduced Cuff-pressure of the Laryngeal Tube Under General Anesthesia
Acronym: LTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, Marc Kriege,MD, Rüdiger Noppens, MD, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGU
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Airway Morbidity
Keywords: laryngeal tube; cuff pressure; leakage; laryngeal mask

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduce Cuff Pressure (Experimental): Cuff Pressure difference between inspiration and expiration is measured.
  Interventions: Device: Reduce Cuff pressure

INTERVENTIONS:
Device: Reduce Cuff pressure — We reduce the Cuff Pressure from the LTS-D (Laryngeal Tube suction) from 60 to 50 to 40 to 30cmH2O and measure the Delta from Inspiration to Expiration Tidalvolume (Delta Vt). The Delta Vt shows the actual leakage.

SUMMARY:
Optimization the cuff pressure of the laryngeal tube (LT) in relation of the mechanical ventilation, and the reduction of potential leakage mucosal trauma. Comparison of the tightness of LT between the filling volume specified by the manufacturer (connectors are color coded syringe and blocker), 60cmH₂O, 50cmH₂O, 40cmH₂Ound 30cmH₂O. The measurement of the leakage occurs in ml / kg body weight.

DETAILED DESCRIPTION:
The ventilation of both cuffs of the laryngeal tube by using the color coding of syringe and connector is a simple, fast and easy way to stabilize the tube and secure seal against the surrounding tissue.

The user of this method has only knowledge of the volume (ml), with which the cuff is vented, but not over the cuff pressure (cmH₂O) itself.

Permanently high pressures can cause to a lesions to necrosis in the adjacent tissue, on the other hand, the material of the bulging cuff fits less well the anatomy of the patient, leading to leaks in the breathing circuit.

Studies of pediatric anesthesia show that on 40cmH₂O reduces the volume of the leak in the laryngeal mask airway by reducing the cuff pressure and the ventilation is improved in sequence.

In the proposed study, the volume of leakage at the fill volume specified by the manufacturer (color coding), 60cmH₂O, 50cmH₂O, 40cmH₂O and 30cmH₂O to be captured.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* No concurrent participation in another study
* capacity to consent
* Present written informed consent of the research participant
* Elective surgery under general anesthesia
* Height> 150cm

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* emergency patients
* Emergency situations in the context of a Difficult Airway Management
* ASA classification> 3
* situations where the possibility of accumulated gastric contents
* Indications for intubation with endotracheal tube
* Height <150cm
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Leakage between the different Cuff Pressure | < 5 Minutes
  We want to measure the tightness of the reduced Cuff Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger Noppens, MD, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Result] Janig C, Marquardt S, Dietze T, Nitsche T. Laryngeal tube placement on manikin by laypersons: is there a possibility for 'public access airway management'? Eur J Emerg Med. 2014 Feb;21(1):65-8. doi: 10.1097/MEJ.0b013e328364a152. PMID 23887642
- [Derived] Kriege M, Alflen C, Eisel J, Ott T, Piepho T, Noppens RR. Evaluation of the optimal cuff volume and cuff pressure of the revised laryngeal tube "LTS-D" in surgical patients. BMC Anesthesiol. 2017 Feb 2;17(1):19. doi: 10.1186/s12871-017-0308-4. PMID 28152975